CLINICAL TRIAL: NCT02395458
Title: Efficacy on Helicobacter Pylori Eradication With Sequential Antibiotic Compared to Triple Therapy for 14 Days
Brief Title: Efficacy on Helicobacter Pylori Eradication With Two Antibiotic Regimens
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Jorge Escobedo de la Pena, Head of the Clinical Research Centre, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2013-3609-22
Record Dates: First submitted 2015-03-12; First posted 2015-03-23 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Helicobacter Infections
Keywords: Sequential therapy; Triple therapy; Eradication
MeSH Terms: conditions — Helicobacter Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sequential therapy (Experimental): Patient receive Omeprazole plus amoxicillin during 5 days and then omeprazole plus clarithromycin and metronidazole during another 5 days
  Interventions: Drug: Sequential therapy
- Triple therapy (Active Comparator): Patient receive Omeprazole plus clarithromycin and amoxicillin during 14 days
  Interventions: Drug: Triple therapy

INTERVENTIONS:
Drug: Sequential therapy — Patient receive Omeprazole plus amoxicillin during 5 days and then omeprazole plus clarithromycin and metronidazole during another 5 days
  Other Names: Omeprazole-Amoxicillin-Clarithromycin-Metronidazole
  Arms: Sequential therapy
Drug: Triple therapy — Patient receive Omeprazole plus amoxicillin and Clarithromycin during 14 days
  Other Names: Omeprazole-Clarithromycin-Metronidazole
  Arms: Triple therapy

SUMMARY:
Clinical trial to compare efficacy on eradicating Helicobacter pylori with two antibiotic strategies: sequential with amoxicillin and omeprazole 5 days and clarithromycin with metronidazole and omeprazole 5 days or omeprazole with clarithromycin and amoxicillin 14 days.

DETAILED DESCRIPTION:
In patients with documented infection with Helicobacter pylori after endoscopy and biopsy, two modalities of treatment were compared, and after a control endoscopy and biopsy, eradication was assessed as well as side effects of both treatments.

ELIGIBILITY:
Inclusion Criteria:

* Helicobacter pylori infection in biopsy
* Eradication required

Exclusion Criteria:

* Antibiotic received two weeks prior
* Previous treatment for H pylori infection
* Allergy to any of the treatment drugs
* Smoking > 5 cigarettes daily.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2013-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Eradication | 6 to 8 week after treatment
  Helicobacter pylori in gastric biopsy

SECONDARY OUTCOMES:
Side effects | two weeks after beginning of treatment
  Nausea, vomiting, stomach ache